CLINICAL TRIAL: NCT06236633
Title: Evaluation of the Safety and Efficacy of Ischemic Preconditioning by Embolization of the Inferior Mesenteric Artery in Oncologic Surgery for Tumors of the Lower and Middle Rectum. Bicentric Exploratory Pilot Study
Brief Title: Safety & Efficacy of Ischemic Preconditioning by Embolization of the Inferior Mesenteric Artery in Surgery for Tumors of Lower and Middle Rectum
Acronym: AMIREMBOL_2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIMAO/2022-1/MB-01
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Cancer, Rectal
Keywords: Ischemic preconditioning surgery; Cancer, Rectal; Inferior Mesenteric Artery Embolus
MeSH Terms: conditions — Rectal Neoplasms | interventions — Ischemic Preconditioning

STUDY DESIGN:
Intervention Model Description: Pilot exploratory descriptive prospective bicentric study to evaluate the safety and efficacy of an innovative procedure: inferior mesenteric artery embolization prior to rectal cancer surgery involving 2 groups: one with standard treatment and the other with inferior mesenteric artery embolization.
Masking Description: Due to the type of intervention and the design of the study, the patient and the referring caregivers cannot be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): In the control group, patients will undergo standard management.
- Ischemic preconditioning group (Experimental): In the experimental group, patients will undergo preoperative arteriography and ischemic preconditioning One blood sample will be taken before and two samples taken after embolization of the IMA.
  These patients will receive a phone call on Day 7 post embolization. A blood sample will also be taken at the time of surgery.
  Interventions: Procedure: Ischemic preconditioning; Procedure: Arteriogram

INTERVENTIONS:
Procedure: Ischemic preconditioning — Embolization performed via a common right femoral or radial approach, depending on the patient's conformation. Minor complications such as hematoma at the puncture site are rare in less than 1% of cases, and serious complications are exceptional. Proximal occlusion of the inferior mesenteric artery, before its dividing branches, using material adapted to arterial occlusion according to anatomical findings. Proximal occlusion during embolization is evaluated by intravascular injection into the inferior mesenteric artery, and resumption of vascularization of the distal inferior mesenteric artery is controlled by the border arcade injecting into the superior mesenteric artery. In the event of a high-risk anatomical variant, or absence of a border arcade, no embolization will be performed and the patient will be excluded from the study; this will represent no more than 1-2% of patients (surgical series describing 0.83% of ischemia in connection with absence of a border arcade).
  Arms: Ischemic preconditioning group
Procedure: Arteriogram — The interventional radiologist performs an arteriogram of the inferior and superior mesenteric arteries (IMA and SMA respectively) to check that the SMA is free of anomalies and that the IMA has a proximal trunk long enough for embolization. The radiologist also checks for the presence of a colonic border arcade. If this is absent, embolization will not be performed: the patient will be excluded from the study.This arteriogram is carried out under local anaesthetic specifically for research purposes, as follows: Common right femoral or radial approach and placement of a small introducer. Selective arteriogram of the inferior and superior mesenteric arteries to check perfusion of the border arcade.Arterial closure system or manual compression. Return to surgery or interventional radiology department. Patient discharged the same day after medical assessment (surgeon or interventional radiologist).Telephone check-up on Day1 (standard management) and Day 7 (added as part of the protocol).
  Arms: Ischemic preconditioning group

SUMMARY:
The present study will investigate the safety of inferior mesenteric artery embolization prior to rectal surgery, according to IDEAL recommendations (Lancet 2009). It aims to assess the safety of endovascular embolization of the inferior mesenteric artery prior to surgery in patients with rectal tumors, and estimate the potential benefits in terms of time to surgery and the occurrence of post-operative fistulas.The study will also assess the impact of subacute ischemia induced by IMA embolization on colonic vasculature remodeling, colonic ischemic suffering, altered hemostasis and initiation of neo-angiogenesis through blood sampling kinetics.The hypothesis is that ischemic preconditioning by inferior mesenteric artery embolization prior to rectal cancer resection surgery is safe and will result in a decrease in acute relative colon ischemia and a reduction in the rate of fistulas and post-surgical complications. Indeed, we believe that the beneficial effects of the ischemic preconditioning of IMA will be due to better blood perfusion of the colon at 3 weeks, which is apparently linked to remodeling and/or the development of collateral vascularization.

DETAILED DESCRIPTION:
Anastomotic fistulas are the main cause of morbidity and mortality in colorectal surgery. They are responsible for septic complications, leading to increased mortality, local recurrence, repeat surgery and impaired sexual, urinary and digestive function. Fistulas are multifactorial; among the causes, colonic vascularization seems to be a major one. Ligation of the inferior mesenteric artery during rectal surgery has been shown to reduce intraoperative colonic perfusion flow. The left colon is then vascularized only by the colonic border arcade, perfused by the superior mesenteric artery. Ischemic pre-conditioning of the arterial network prior to surgery should ensure better vascularization by developing arterial collaterality and increasing perfusion flow in the colonic border arcade. In view of major advances in interventional radiology, this preconditioning could be achieved by endovascular ligation of the inferior mesenteric artery (IMA), based on the same principle as during surgery: proximal occlusion of the inferior mesenteric artery (IMA), using embolization material (plug or coils), 3 weeks before surgery, to allow the colonic border arcade to develop. We carried out a single-center pilot study (AMIREMBOL 1, NIMAO 2017; Frandon et al. 2022) to assess the feasibility of ischemic preconditioning of the colon for patients with rectal or sigmoid cancer. The study included 10 patients, randomized into two groups: the control group, with preoperative arteriography and standard management and the "embolization" group, with embolization of the IMA three weeks prior to surgery. IMA embolization was successfully performed in all 5 patients in the embolization group, with no major complications. The effect on colonic perfusion, measured by intraoperative Doppler directly on the border arch, with recording of resistance indexes (independent of measurement angle), showed a drop in resistance indexes in the control arm, after ligation of the IMA, which persisted after 5 minutes. In the "Embolization" arm, no drop in this index was reported during surgery, reflecting good development of vascular collaterality and at least relative acute ischemia of the colon after IMA ligation during surgery. Finally, in the "control" group, one anastomotic fistula was reported after surgery and required re-operation. There were no fistulas in the embolization group.

The present study (AMIREMBOL 2) will investigate the safety of IMA embolization prior to rectal surgery, according to IDEAL recommendations (Lancet 2009). Its aim is to assess the safety of endovascular embolization of the IMA prior to surgery in patients with rectal tumors, and to estimate the potential benefits in terms of time to surgery and the occurrence of post-operative fistulas.

The study will also assess the impact of subacute ischemia induced by IMA embolization on colonic vasculature remodeling, colonic ischemic suffering, altered hemostasis and initiation of neo-angiogenesis through blood sampling kinetics.

The hypothesis is that ischemic preconditioning by inferior mesenteric artery (IMA) embolization prior to rectal cancer resection surgery is safe and will result in a decrease in acute relative colon ischemia and a reduction in the rate of fistulas and post-surgical complications. The hypothesis is that the beneficial effects of the ischemic preconditioning of IMA will be due to better blood perfusion of the colon at 3 weeks, which is apparently linked to remodeling and/or the development of collateral vascularization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rectal cancer eligible for surgery with ligation at the origin of the inferior mesenteric artery.
* Patients with free, informed consent.
* Patients affiliated to or benefiting from a health insurance plan.

Exclusion Criteria:

* Patients with a history of colon cancer who has undergone colon resection surgery
* Patients with occlusion of the superior mesenteric artery or stenosis of more than 50%, visible on the CT scan performed as part of conventional management during extension workup.
* Patients with occlusion of the IMA on the extension scan.
* Patients with a systemic disorder responsible for haemostasis (haemophilia, Willebrand's disease, thrombocytopenia) and on anticoagulant therapy.
* Patients taking corticosteroids or immunosuppressants leading to an unacceptable surgical risk.
* Patients with renal insufficiency with clearance < 30mL/min.
* Patients with an allergy to iodine.
* Patients who has had treatment of the abdominal aorta or its branches.
* Patients participating in an interventional study.
* Patients in an exclusion period determined by another study.
* Patients under court protection, guardianship or curatorship.
* Patients unable to give consent.
* Patients for whom it is impossible to provide informed information.
* Pregnant or breast-feeding patients.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Safety of endovascular inferior mesenteric artery embolisation prior to surgical resection of the rectum in patients with tumours of the lower and middle rectum. | Day 7 post embolization (performed 3 weeks before surgical resection of the rectum)
  Percentage of patients with a complication (any grade) within 7 days after embolisation of the inferior mesenteric artery according to the classification of the International Society of Interventional Radiology assessed during the follow-up telephone consultation by the interventional radiologist.
  Complications will be classified as minor (Grades A and B) or Major (grades C to F).
  Grade A = No therapy, no consequence Grade B = Nominal therapy, no consequence. Includes overnight admission for observation only Grade C = Requires therapy, minor hospitalization (<48 hours) Grade D = Requires major therapy. Unplanned increase in level of care. Prolonged hospitalization (>48 hours) Grade E = Permanent adverse sequelae Grade F= Death

SECONDARY OUTCOMES:
Technical success of the embolization procedure | Day 0, on the day of embolization
  A control arteriogram of the inferior and superior mesenteric arteries will be carried out at the end of the embolisation procedure: intravascular injection into the inferior mesenteric artery and control of the resumption of vascularisation of the distal inferior mesenteric artery by the border arcade by injecting into the superior mesenteric artery.
  If embolisation fails, the patient will continue the study.
  The number of failures will be converted into a percentage
Post-surgical complications up to 30 days after surgery. Clavien-Dindo Grade I | Post-operative Day 30
  Percentage of patients presenting a post-operative complication according to the Clavien-Dindo Classification within 30 days of rectal surgery, assessed during hospitalization and at the 1-month post-surgical consultation, according to standard management.
  The Clavien-Dindo classification (Dindo et al 2004, Dindo D. 2004) classifies surgical complications into 7 categories (I, II, IIIa, IIIb, IVa, IVb and V)
Post-surgical complications up to 30 days after surgery. Clavien-Dindo Grade II | Post-operative Day 30
  Percentage of patients presenting a post-operative complication according to the Clavien-Dindo Classification within 30 days of rectal surgery, assessed during hospitalization and at the 1-month post-surgical consultation, according to standard management.
  The Clavien-Dindo classification (Dindo et al 2004, Dindo D. 2004) classifies surgical complications into 7 categories (I, II, IIIa, IIIb, IVa, IVb and V)
Post-surgical complications up to 30 days after surgery. Clavien-Dindo Grade IIIa | Post-operative Day 30
  Percentage of patients presenting a post-operative complication according to the Clavien-Dindo Classification within 30 days of rectal surgery, assessed during hospitalization and at the 1-month post-surgical consultation, according to standard management.
  The Clavien-Dindo classification (Dindo et al 2004, Dindo D. 2004) classifies surgical complications into 7 categories (I, II, IIIa, IIIb, IVa, IVb and V)
Post-surgical complications up to 30 days after surgery. Clavien-Dindo Grade IIIb | Post-operative Day 30
  Percentage of patients presenting a post-operative complication according to the Clavien-Dindo Classification within 30 days of rectal surgery, assessed during hospitalization and at the 1-month post-surgical consultation, according to standard management.
  The Clavien-Dindo classification (Dindo et al 2004, Dindo D. 2004) classifies surgical complications into 7 categories (I, II, IIIa, IIIb, IVa, IVb and V)
Post-surgical complications up to 30 days after surgery. Clavien-Dindo Grade IVa | Post-operative Day 30
  Percentage of patients presenting a post-operative complication according to the Clavien-Dindo Classification within 30 days of rectal surgery, assessed during hospitalization and at the 1-month post-surgical consultation, according to standard management.
  The Clavien-Dindo classification (Dindo et al 2004, Dindo D. 2004) classifies surgical complications into 7 categories (I, II, IIIa, IIIb, IVa, IVb and V)
Post-surgical complications up to 30 days after surgery. Clavien-Dindo Grade IVb | Post-operative Day 30
  Percentage of patients presenting a post-operative complication according to the Clavien-Dindo Classification within 30 days of rectal surgery, assessed during hospitalization and at the 1-month post-surgical consultation, according to standard management.
  The Clavien-Dindo classification (Dindo et al 2004, Dindo D. 2004) classifies surgical complications into 7 categories (I, II, IIIa, IIIb, IVa, IVb and V)
Post-surgical complications up to 30 days after surgery. Clavien-Dindo Grade V | Post-operative Day 30
  Percentage of patients presenting a post-operative complication according to the Clavien-Dindo Classification within 30 days of rectal surgery, assessed during hospitalization and at the 1-month post-surgical consultation, according to standard management.
  The Clavien-Dindo classification (Dindo et al 2004, Dindo D. 2004) classifies surgical complications into 7 categories (I, II, IIIa, IIIb, IVa, IVb and V)
Rate of fistulas up to 30 days after surgery | Day 0
  Percentage of patients with a fistula within 30 days of rectal surgery, assessed during hospitalization and at the 1-month post-surgical consultation, according to standard management.A fistula will be identified either on the basis of clinical criteria (presence of pus or enteric contents in the drains, leakage of contrast medium through the anastomosis, anastomotic dehiscence during a repeat operation), or on the basis of radiological criteria (presence of an abdominal or pelvic collection in the area of the anastomosis on CT scan) if there is clinical doubt or if a CT scan is carried out for another reason (before stoma closure, for example).
Rate of fistulas up to 30 days after surgery | Post-operative Day 30
  Percentage of patients with a fistula within 30 days of rectal surgery, assessed during hospitalization and at the 1-month post-surgical consultation, according to standard management.A fistula will be identified either on the basis of clinical criteria (presence of pus or enteric contents in the drains, leakage of contrast medium through the anastomosis, anastomotic dehiscence during a repeat operation), or on the basis of radiological criteria (presence of an abdominal or pelvic collection in the area of the anastomosis on CT scan) if there is clinical doubt or if a CT scan is carried out for another reason (before stoma closure, for example).
Duration of post-surgical hospitalization | Up to 30 days after rectal surgery
  Length of hospital stay (number of days)
Degree of difficulty experienced by the visceral surgeon during surgery | Week 3 to 4 on the day of rectal surgery
  Surgeon's assessment of degree of difficulty using a 4-point Likert scale after each operation as follows :
  1= Dissection of the inferior mesenteric artery was standard 2 = Dissection of the inferior mesenteric artery was more complicated than expected 3 = Dissection of the inferior mesenteric artery was much more complicated than expected; 4 = Dissection of the inferior mesenteric artery was Very difficult.
Systemic inflammation markers: Pro-inflammation cytokines | Day 0 (on the day of inclusion)
  Pro-inflammation cytokines (IL-1β, IL-6, IL-8, Tumor Necrosis Factor-α and Interferon-ɣ) will be measured as percentages
Systemic inflammation markers: Pro-inflammation cytokines | 25 minutes before embolization
  Pro-inflammation cytokines (IL-1β, IL-6, IL-8, Tumor Necrosis Factor-α and Interferon-ɣ) will be measured as percentages
Systemic inflammation markers: Pro-inflammation cytokines | 60 minutes after embolization
  Pro-inflammation cytokines (IL-1β, IL-6, IL-8, Tumor Necrosis Factor-α and Interferon-ɣ) will be measured as percentages
Systemic inflammation markers: Pro-inflammation cytokines | Week 3 to 4 after patient induction just before rectal surgery
  Pro-inflammation cytokines (IL-1β, IL-6, IL-8, Tumor Necrosis Factor-α and Interferon-ɣ) will be measured as percentages
Systemic inflammation markers: Complement protein C3 | Day 0 (on the day of inclusion)
  Complement protein C3 will be measured as a percentage
Systemic inflammation markers: Complement protein C3 | 25 minutes before embolization
  Complement protein C3 will be measured as a percentage
Systemic inflammation markers: Complement protein C3 | 60 minutes after embolization
  Complement protein C3 will be measured as a percentage
Systemic inflammation markers: Complement protein C3 | Week 3 to 4 after patient induction just before rectal surgery
  Complement protein C3 will be measured as a percentage
Anti-inflammation markers: | Day 0 (on the day of inclusion)
  IL-10 and Transforming Growth Factor-β will be measured as percentages
Anti-inflammation markers: | 25 minutes before embolization
  IL-10 and Transforming Growth Factor-β will be measured as percentages
Anti-inflammation markers: | 60 minutes after embolization
  IL-10 and Transforming Growth Factor-β will be measured as percentages
Anti-inflammation markers: | Week 3 to 4 after patient induction just before rectal surgery
  IL-10 and Transforming Growth Factor-β will be measured as percentages
Hemostasis markers : Von Willebrand factor | Day 0 (on the day of inclusion)
  Von Willebrand factor will be measured.
Hemostasis markers : Von Willebrand factor | 25 minutes before embolization
  Von Willebrand factor will be measured.
Hemostasis markers : Von Willebrand factor | 60 minutes after embolization
  Von Willebrand factor will be measured.
Hemostasis markers : Von Willebrand factor | Week 3 to 4 after patient induction just before rectal surgery
  Von Willebrand factor will be measured.
Hemostasis markers : coagulation factor V | Day 0 (on the day of inclusion)
  Coagulation factor V will be measured.
Hemostasis markers : coagulation factor V | 25 minutes before embolization
  Coagulation factor V will be measured.
Hemostasis markers : coagulation factor V | 60 minutes after embolization
  Coagulation factor V will be measured.
Hemostasis markers : coagulation factor V | Week 3 to 4 after patient induction just before rectal surgery
  Coagulation factor V will be measured.
Hemostasis markers : D-dimers | Day 0 (on the day of inclusion)
  D-dimers will be measured
Hemostasis markers : D-dimers | 25 minutes before embolization
  D-dimers will be measured
Hemostasis markers : D-dimers | 60 minutes after embolization
  D-dimers will be measured
Hemostasis markers : D-dimers | Week 3 to 4 after patient induction just before rectal surgery
  D-dimers will be measured
Hemostasis markers : platelet-activating factor (PAF) | Day 0 (on the day of inclusion)
  Platelet-activating factor (PAF) will be measured
Hemostasis markers : platelet-activating factor (PAF) | 25 minutes before embolization
  Platelet-activating factor (PAF) will be measured
Hemostasis markers : platelet-activating factor (PAF) | 60 minutes after embolization
  Platelet-activating factor (PAF) will be measured
Hemostasis markers : platelet-activating factor (PAF) | Week 3 to 4 after patient induction just before rectal surgery
  Platelet-activating factor (PAF) will be measured
Hemostasis markers : prostaglandin E4 | Day 0 (on the day of inclusion)
  Prostaglandin E4 will be measured
Hemostasis markers : prostaglandin E4 | 25 minutes before embolization
  Prostaglandin E4 will be measured
Hemostasis markers : prostaglandin E4 | 60 minutes after embolization
  Prostaglandin E4 will be measured
Hemostasis markers : prostaglandin E4 | Week 3 to 4 after patient induction just before rectal surgery
  Prostaglandin E4 will be measured
Hemostasis markers : Thromboxane B2 | Day 0 (on the day of inclusion)
  Thromboxane B2 will be measured.
Hemostasis markers : Thromboxane B2 | 25 minutes before embolization
  Thromboxane B2 will be measured.
Hemostasis markers : Thromboxane B2 | 60 minutes after embolization
  Thromboxane B2 will be measured.
Hemostasis markers : Thromboxane B2 | Week 3 to 4 after patient induction just before rectal surgery
  Thromboxane B2 will be measured.
Markers of tissue inflammation: Blood pH | Day 0 (on the day of inclusion)
  Blood pH will be measured
Markers of tissue inflammation: Blood pH | 25 minutes before embolization
  Blood pH will be measured
Markers of tissue inflammation: Blood pH | 60 minutes after embolization
  Blood pH will be measured
Markers of tissue inflammation: Blood pH | Week 3 to 4 after patient induction just before rectal surgery
  Blood pH will be measured
Markers of tissue inflammation: ischemia-modified albumin | Day 0 (on the day of inclusion)
  Ischemia-modified albumin will be measured
Markers of tissue inflammation: ischemia-modified albumin | 25 minutes before embolization
  Ischemia-modified albumin will be measured
Markers of tissue inflammation: ischemia-modified albumin | 60 minutes after embolization
  Ischemia-modified albumin will be measured
Markers of tissue inflammation: ischemia-modified albumin | Week 3 to 4 after patient induction just before rectal surgery
  Ischemia-modified albumin will be measured
Markers of tissue inflammation:intestinal fatty acid-binding protein (I-FABP) | Day 0 (on the day of inclusion)
  intestinal fatty acid-binding protein (I-FABP) will be measured
Markers of tissue inflammation:intestinal fatty acid-binding protein (I-FABP) | 25 minutes before embolization
  intestinal fatty acid-binding protein (I-FABP) will be measured
Markers of tissue inflammation:intestinal fatty acid-binding protein (I-FABP) | 60 minutes after embolization
  intestinal fatty acid-binding protein (I-FABP) will be measured
Markers of tissue inflammation:intestinal fatty acid-binding protein (I-FABP) | Week 3 to 4 after patient induction just before rectal surgery
  intestinal fatty acid-binding protein (I-FABP) will be measured
Markers of tissue inflammation: L-lactate | Day 0 (on the day of inclusion)
  L-lactate will be measured
Markers of tissue inflammation: L-lactate | 25 minutes before embolization
  L-lactate will be measured
Markers of tissue inflammation: L-lactate | 60 minutes after embolization
  L-lactate will be measured
Markers of tissue inflammation: L-lactate | Week 3 to 4 after patient induction just before rectal surgery
  L-lactate will be measured
Markers of tissue inflammation: D-lactate | Day 0 (on the day of inclusion)
  D-lactate will be measured
Markers of tissue inflammation: D-lactate | 25 minutes before embolization
  D-lactate will be measured
Markers of tissue inflammation: D-lactate | 60 minutes after embolization
  D-lactate will be measured
Markers of tissue inflammation: D-lactate | Week 3 to 4 after patient induction just before rectal surgery
  D-lactate will be measured
Markers of tissue inflammation: Lactate dehydrogenase | Day 0 (on the day of inclusion)
  Lactate dehydrogenase will be measured
Markers of tissue inflammation: Lactate dehydrogenase | 25 minutes before embolization
  Lactate dehydrogenase will be measured
Markers of tissue inflammation: Lactate dehydrogenase | 60 minutes after embolization
  Lactate dehydrogenase will be measured
Markers of tissue inflammation: Lactate dehydrogenase | Week 3 to 4 after patient induction just before rectal surgery
  Lactate dehydrogenase will be measured
Markers of neoangiogenesis : CD34 | Day 0 (on the day of inclusion)
  CD34 will be measured
Markers of neoangiogenesis : CD34 | 25 minutes before embolization
  CD34 will be measured
Markers of neoangiogenesis : CD34 | 60 minutes after embolization
  CD34 will be measured
Markers of neoangiogenesis : CD34 | Week 3 to 4 after patient induction just before rectal surgery
  CD34 will be measured
Markers of neoangiogenesis : transcription factor HIF1-α | Day 0 (on the day of inclusion)
  Transcription factor HIF1-α will be measured
Markers of neoangiogenesis : transcription factor HIF1-α | 25 minutes before embolization
  Transcription factor HIF1-α will be measured
Markers of neoangiogenesis : transcription factor HIF1-α | 60 minutes after embolization
  Transcription factor HIF1-α will be measured
Markers of neoangiogenesis : transcription factor HIF1-α | Week 3 to 4 after patient induction just before rectal surgery
  Transcription factor HIF1-α will be measured
Markers of neoangiogenesis : Growth factors | Day 0 (on the day of inclusion)
  Growth factors and their receptors, notably vascular endothelial growth factor (VEGF) and vascular endothelial growth factor receptor (VEGFR), fibroblast growth factor (FGF) and fibroblast growth factor receptor (FGFR) and platelet-derived growth factor (PDGF) and platelet-derived growth factor receptor (PDGFR) will be measured
Markers of neoangiogenesis : Growth factors | 25 minutes before embolization
  Growth factors and their receptors, notably vascular endothelial growth factor (VEGF) and vascular endothelial growth factor receptor (VEGFR), fibroblast growth factor (FGF) and fibroblast growth factor receptor (FGFR) and platelet-derived growth factor (PDGF) and platelet-derived growth factor receptor (PDGFR) will be measured
Markers of neoangiogenesis : Growth factors | 60 minutes after embolization
  Growth factors and their receptors, notably vascular endothelial growth factor (VEGF) and vascular endothelial growth factor receptor (VEGFR), fibroblast growth factor (FGF) and fibroblast growth factor receptor (FGFR) and platelet-derived growth factor (PDGF) and platelet-derived growth factor receptor (PDGFR) will be measured
Markers of neoangiogenesis : Growth factors | Week 3 to 4 after patient induction just before rectal surgery
  Growth factors and their receptors, notably vascular endothelial growth factor (VEGF) and vascular endothelial growth factor receptor (VEGFR), fibroblast growth factor (FGF) and fibroblast growth factor receptor (FGFR) and platelet-derived growth factor (PDGF) and platelet-derived growth factor receptor (PDGFR) will be measured
Markers of epithelial-mesenchymal transition : matrix metallo-protease - 2 | Day 0 (on the day of inclusion)
  Matrix metallo-protease - 2 will be measured
Markers of epithelial-mesenchymal transition : matrix metallo-protease - 2 | 25 minutes before embolization
  Matrix metallo-protease - 2 will be measured
Markers of epithelial-mesenchymal transition : matrix metallo-protease - 2 | 60 minutes after embolization
  Matrix metallo-protease - 2 will be measured
Markers of epithelial-mesenchymal transition : matrix metallo-protease - 2 | Week 3 to 4 after patient induction just before rectal surgery
  Matrix metallo-protease - 2 will be measured
Markers of epithelial-mesenchymal transition : matrix metallo-protease - 9 | Day 0 (on the day of inclusion)
  Matrix metallo-protease - 9 will be measured
Markers of epithelial-mesenchymal transition : matrix metallo-protease - 9 | 25 minutes before embolization
  Matrix metallo-protease - 9 will be measured
Markers of epithelial-mesenchymal transition : matrix metallo-protease - 9 | 60 minutes after embolization
  Matrix metallo-protease - 9 will be measured
Markers of epithelial-mesenchymal transition : matrix metallo-protease - 9 | Week 3 to 4 after patient induction just before rectal surgery
  Matrix metallo-protease - 9 will be measured
Markers of epithelial-mesenchymal transition : transcription factors | Day 0 (on the day of inclusion)
  Transcription factors SNAI2 (SLUG), SNAI1 (SNAIL) and zinc-finger E-box binding homeobox (ZEB-1) will be measured
Markers of epithelial-mesenchymal transition : transcription factors | 25 minutes before embolization
  Transcription factors SNAI2 (SLUG), SNAI1 (SNAIL) and zinc-finger E-box binding homeobox (ZEB-1) will be measured
Markers of epithelial-mesenchymal transition : transcription factors | 60 minutes after embolization
  Transcription factors SNAI2 (SLUG), SNAIL (SNAI1) and zinc-finger E-box binding homeobox (ZEB-1) will be measured
Markers of epithelial-mesenchymal transition : transcription factors | Week 3 to 4 after patient induction just before rectal surgery
  Transcription factors SNAI2 (SLUG), SNAIL (SNAI1) and zinc-finger E-box binding homeobox (ZEB-1) will be measured

OTHER OUTCOMES:
Gender | Day 0, on the day of inclusion
  Male/Female
Age | Day 0, on the day of inclusion
  In years
Height | Day 0, on the day of inclusion
  In centimeters
Tumor stage | Day 0, on the day of inclusion
  Stage 0: Cancer cells are limited to the surface of the rectal lining. Stage I: Tumor has grown below the lining and possibly into the rectal wall. Stage II: Tumor has grown into the rectal wall and might extend into tissues around the rectum.
  Stage III: Tumor has invaded the lymph nodes next to the rectum and some tissues outside of the rectal wall.
  Stage IV: Cancer has spread to distant organs, such as the liver or lungs.
Tumor, Node and Metastasis staging (TNM) | Day 0, on the day of inclusion
  Tis:tumor in situ, only in mucosa.T1:tumor only in inner layer of bowel T2:tumor in muscle layer of the bowel wall T3:tumor in outer lining of bowel wall but not through it. T4a: tumor has gone through outer lining of bowel wall and into the peritoneum. T4b:tumor has grown through the bowel wall into nearby organs. N:cancer spread to lymph nodes? N0: no lymph nodes containing cancer cells. N1a:cancer cells in 1 nearby lymph node, N1b:cancer cells in 2 or 3 nearby lymph nodes,N1c:nearby lymph nodes do not contain cancer, but cancer cells in the tissue near the tumor. N2a:cancer cells in 4 to 6 nearby lymph nodes, N2b:cancer cells in >7 nearby lymph nodes. M:cancer in another part of the body (metastasis)? M0:cancer not spread to other organs, M1:cancer spread to elsewhere in the body. M1a: cancer spread to 1 distant site or organ, e.g. liver, but not to peritoneum, M1b:cancer spread to >2 distant sites, not to tissue lining the peritoneum M1c:cancer in distant organs and peritoneum.
Circumferential resection margin | Week 3 or 4 on the day of surgery
  In millimeters
Distance from the lower pole of the tumor relative to the upper edge of the anal sphincter | Week 3 or 4 on the day of surgery
  In millimeters
Bi-ischial diameter | Week 3 or 4 on the day of surgery
  In millimeters
Bi-uterine diameter | Week 3 or 4 on the day of surgery
  In millimeters
Mesorectal area | Week 3 or 4 on the day of surgery
  In square millimeters
Type of surgery | Week 3 or 4 on the day of surgery
  * Colorectal or anal anastomosis
  * Mechanical or manual surgery
  * Intersphincteric dissection Yes/ No, partial or total
  * Delayed colo-anal anastomosis.
Cardiovascular risk factors | Day 0 on the day of inclusion
  All cardiovascular risk factors will be recorded
Presence of the border arcade, occlusion of the mesenteric artery during arteriography. | Day 0 on the day of inclusion
  YES/NO
Operative data | Week 3 or 4 on the day of surgery
  Operative data: mobilisation of the colonic angle and ligation of the mesenteric vein.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Saint-Eloi, Montpellier
  - Institut du Cancer de Montpellier, Montpellier
  - CHU de Nîmes, Nîmes